CLINICAL TRIAL: NCT03518281
Title: A Single Center, Randomized, Double-blind, Placebo-controlled, Parallel Study to Investigate the Ability of a Euglena Beta Glucan Supplementation to Augment Immune Function in Endurance Athletes
Brief Title: Ability of a Euglena Beta Glucan Supplementation to Augment Immune Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kemin Foods LC (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 18ECHK-1
Record Dates: First submitted 2018-01-31; First posted 2018-05-08 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-01

CONDITIONS: Symptoms Flu; Symptoms Cold

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All parties, except an outside person not involved in the study, will be blinded to the treatment conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Treatment (Experimental): Whole Cell Euglena delivering βeta Glucan
  Interventions: Dietary Supplement: Whole Cell Euglena containing Beta Glucan

INTERVENTIONS:
Dietary Supplement: Whole Cell Euglena containing Beta Glucan — Whole Cell Euglena containing >50% Beta Glucan
  Arms: Treatment
Dietary Supplement: Placebo — microcrystalline cellulose, hypromellose, titanium dioxide, water
  Arms: Placebo

SUMMARY:
Upper respiratory tract infections cause cold and flu-like symptoms and are the most common form of acute illness. Certain populations are at increased risk of upper respiratory tract infections including athletes who train at a high level of intensity for prolonged periods of time. Consequently, some athletes experience higher rates of cold and flu-like symptoms than the general population.

Euglena gracilis is a micro-algae which can synthesize many nutrients necessary for human health, including insoluble beta glucan. Thus, intake of whole cell Euglena may be beneficial to athletes by providing essential vitamins to optimize immune function.

DETAILED DESCRIPTION:
At screening, an informed consent form will be given to the potential volunteer. They will be required to read the information and be given the opportunity to seek more information if needed, or provided with the option of taking the consent form home to review prior to making their decision. If agreeable, the volunteer will sign the consent form and receive a duplicate of the signed copy. Once consent has been obtained, the screening visit will proceed.

Screening assessments include:

1. Review of medical history, concomitant therapies and current health status (weight, height, BMI, vital signs, safety blood work)
2. Assesses inclusion and exclusion criteria
3. Urine pregnancy test for female potential participants that are not post-menopausal

Eligible participants will return to the clinic for baseline assessments. Baseline (day 0) assessments include:

1. Review of concomitant therapies and current health status
2. Review pre-supplement emergent AEs
3. Reassess inclusion and exclusion criteria
4. Randomization of eligible participants
5. Dispense daily upper respiratory tract symptom questionnaire
6. Collect saliva sample for measurement of secretory IgA
7. Collect blood sample for the analysis of cell activity
8. Administer mood and stress questionnaire in-clinic
9. Dispense daily gastrointestinal and bowel questionnaire
10. Dispense investigational product and instruct participants on use
11. Dispense daily study diary

At the end-of-study visit (Day 90) participants will return to the clinic for Visit 3 assessments with unused investigational product, completed study diaries, daily symptom questionnaires, daily gastrointestinal and bowel diaries.

Visit 3 assessments include:

1. Collection of all study diaries
2. Return of unused investigational product and calculate compliance
3. Review of concomitant therapies and adverse events
4. Check of health status (vitals, BMI, safety bloodwork)
5. Administer mood and stress questionnaire in-clinic.
6. Collect saliva sample for an end-of-study measurement of secretory IgA
7. Complete Product Tolerability and Perception Questionnaire

ELIGIBILITY:
Inclusion Criteria:

1. Body Mass Index (BMI) > 18 kg/m2 to <35 kg/m2.
2. Willing to comply with a wash-out period for nutritional supplements known to affect immune function and to not consume these supplements for the entire study period
3. Females of childbearing potential must agree to use a medically approved method of birth control
4. Agree to maintaining a consistent diet and lifestyle routine throughout the study
5. An endurance training athlete
6. Healthy as determined by laboratory results and medical history

Exclusion Criteria:

1. Women who are pregnant, breastfeeding, or planning to become pregnant during the course of the trial
2. Verbal confirmation of previous major gastrointestinal surgery
3. Consuming doses of beta-glucan-containing nutritional supplements
4. Chronic consumption of anti-inflammatory medications
5. Taking antibiotics within 4 weeks of screening and during the study period
6. Verbal confirmation of a diagnosed chronic inflammatory condition or autoimmune disorder
7. Verbal confirmation of Type I or Type II diabetes or clinically important renal, hepatic, cardiac, pulmonary, pancreatic, neurologic, or biliary disorder, or a recent history (prior 2 years) of cancer other than non-melanoma skin cancer
8. Currently taking antipsychotic medications
9. Chronic recurring respiratory signs and symptoms due to allergies (including seasonal allergies) or chronic bronchitis, asthma, or wheezing
10. Use of immunomodulators (including corticosteroids) such as immunosuppressant or immunostimulant medications within 4 weeks of baseline and during the study period
11. Chronic use of Antacids and Proton Pump Inhibitors (PPI)
12. Individuals who have received or are planning to receive the flu vaccination for the current flu season
13. Active infection or signs/symptoms of an acute infection
14. Heavy use of tobacco
15. Alcohol or drug abuse within the last 2 years

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Incidence of upper respiratory tract infections | ANOVA of 90 day supplementation
  incidence of very mild/mild/ moderate/ severe upper respiratory tract infection symptoms

SECONDARY OUTCOMES:
Symptom Duration | 30 and 90 days
  Duration of very mild/mild/moderate/sever upper respiratory tract infection symptoms
Stress | 90 days
  Effect of treatment on Stress via Perceived Stress Scale Total Score
Secretory IgA | 90 days
  Effect of treatment on secretory IgA levels
Natural Killer (NK) Cell Population | 90 days
  Effect of treatment on NK cell population changes
Gastrointestinal status | 30 and 90 days
  Effect of treatment on gastrointestinal status via questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- KGK Science Inc., London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No